CLINICAL TRIAL: NCT06395766
Title: Assessment of Quality of Life and Social Support Gained in Patients Before and After Laparoscopic Surgery for Cancer of the Rectum and Cancer of the Right Part of the Intestine (Cecum, Ascending Colon)
Brief Title: Assessment of Quality of Life and Social Support Gained in Patients Before and After Colorectal Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Edyta Laska, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: 30/2023
Record Dates: First submitted 2024-01-01; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BREF,MSPSS — 1. abbreviated version of the quality of life assessment questionnaire - The World Health Organization Quality of Life (WHOQOL )
  2. the Zimet Multidimensional Scale of Perceived Social Support -. The original version on the MSPSS

SUMMARY:
* evaluation of the quality of life of patients before and after laparoscopic surgery for rectal cancer and cancer of the right part of the intestine at different stages of the disease, whether it depends on the size of the tumor, neoadjuvant treatment, type of cancer and its location
* Multidimensional assessment of perceived social support (considering three sources of support: significant person, family and friends) of patients before and after laparoscopic surgery for rectal cancer and cancer of the right part of the intestine, whether it depends on the stage of the disease, the location of the tumor lesion and the treatment undertaken

DETAILED DESCRIPTION:
Specific scientific objectives:

* To evaluate the quality of life of patients before and after laparoscopic surgery for rectal cancer and right-sided colon cancer at different stages of disease, whether it depends on tumor size, neoadjuvant treatment, type of cancer and its location
* Multidimensional evaluation of perceived social support (considering three sources of support: significant person, family and friends) of patients before and after laparoscopic surgery for rectal cancer and cancer of the right part of the intestine, whether it depends on the stage of the disease, the location of the tumor lesion and the treatment undertaken

Scientific (research) problems:

* What is the quality of life of patients before surgery, and what is the quality of life after laparoscopic surgery for rectal cancer and cancer of the right side of the intestine at different stages of oncological disease? Does quality of life depend on the size of the tumor, location, advancement or type of treatment undertaken?
* How do patients rate the received social support both before and after laparoscopic surgery for rectal cancer and right colon cancer ?
* Did the obtained social support in the patient at each stage of the disease ( before surgery, after surgery) depend on the advancement of the oncological lesion, the location of the tumor lesion and the treatment undertaken ? 2 Methodology of the study The study will be carried out at the General Surgery Clinical Department of the John Grande Hospital of the Order of St. John of God in Krakow after obtaining permission from the facility's management.

Each patient qualified for laparoscopic surgery for rectal cancer and cancer of the right side of the intestine who simultaneously agreed to participate in the study anonymously was included in the study group.

ELIGIBILITY:
Inclusion criteria for the study:

* clinical diagnosis of rectal cancer and right colon cancer
* laparoscopic surgery

Study exclusion criteria:

- surgery by traditional method

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each patient who is admitted to the surgical ward with a diagnosis of rectal cancer and cancer of the right side of the intestine and is qualified for laparoscopic surgery will receive written consent for the study and the processing of personal data, as well as information for the researcher with questionnaires, and then if he or she agrees in writing will be recruited for the study. The patient's personal data processing information will be retained for the study until its completion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed using The World Health Organization Quality of Life (WHOQOL) scale.Social support assessed using Zimet's Multidimensional Perceived Social Support Scale - the original version on the MSPSS. | 12 months to 24 months
  Quality of life assessed using The World Health Organization Quality of Life (WHOQOL-BREF) scale questionnaire which contains 26 questions analyzing four domains of life and separately perception of quality of life and self-assessment of health status.
  It is used to assess the quality of life of both healthy and sick people in clinical practice and addresses the following domains of quality of life: somatic functioning, psychological functioning, social functioning and community functioning.
  Social support assessed using Zimet's Multidimensional Perceived Social Support Scale - the original version on the MSPSS.
  The Multidimensional Scale of Perceived Social Support takes into account the multidimensionality of perceived social support, considering three primary sources of support: significant other, family and friends. The scale consists of 12 statements, which the subject addresses using a seven-point Likert scale, where 1 means "strongly disagree" and 7 means "strongly agree."

CONTACTS AND LOCATIONS:
Locations (1):
- John Grande Hospital of the Monastery of St. John of God, Krakow, Lesserpoland, Poland

IPD SHARING:
Plan to Share IPD: No